CLINICAL TRIAL: NCT01561196
Title: Conventional vs. Ultrasound Guided Arteria Cannulation, With and Without Local Anesthesia
Brief Title: Conventional Verses Ultrasound Guided Arteria Cannulation, With and Without Local Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marlene A Hansen, Stud.med (Other)
Responsible Party: Sponsor-Investigator, Marlene A Hansen, Stud.med, stud.med, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Sloth1
Record Dates: First submitted 2012-03-13; First posted 2012-03-22 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Heart Disease
Keywords: arteria cannulation; Ultrasound; pain; complications
MeSH Terms: conditions — Heart Diseases; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound guided arterial cannulation (Active Comparator): The arterial needle is placed using ultrasound monitoring for guiding the operator.
  Interventions: Procedure: arterial catheterisation
- Conventional cannulation (Active Comparator): the arterial needle is placed using the traditional method and lidocaine. The operator decides where to place the needle in the forearm
  Interventions: Procedure: arterial catheterisation

INTERVENTIONS:
Procedure: arterial catheterisation — arterial catheterisation in Arterial Radialis
  Other Names: ICD10 I95.9

SUMMARY:
The aim of the project is to compare two methods for arterial cannulation. The traditional method with ultrasound guided cannulation. The investigators goal is to improve this procedure to reduce pain and complications.

DETAILED DESCRIPTION:
The practice of placing vascular catheters is used many times every day at almost every hospital. It is a safe procedure which generally does not imply problems. Though the procedural optimum aren't reached. The procedure still fails some times and induce complications. When the catheter is placed using the traditional method the pulse is palpated by the operator's fingers. This is only to be done near the hand wrist. In this position the catheter steadiness is fragile but because the pulse can't be sensed more proximal the operator is forced to choose this position. This it though a problem that can be solved by non invasive visualization technology. Ultrasound-guidance for central vascular access is already well-established. However, in recent years ultrasound-guidance for peripheral vascular access has gained popularity too. The evidence of multiple studies demonstrates increased success rate and reduced complication rate with ultrasound compared to blind landmark technique for vascular catheter placement.

In recent years there have been both procedural technique and technology improvements in the field of ultrasound. This has led to the improvement of procedural catheterisation techniques that now can be done by novices with higher attempt success rate than traditional method. One technique that is gaining success is the short-axis-out-of-plane technique (SAX-OOP) with dynamic-needle-tip-tracking (DNTT).Using the ultrasound machine the needle can be placed in a more proximal direction on the forearm and the investigators believe that by the help of the exposed procedure on the monitor many complications can be reduced.

Hypothesis; Firstly the investigators hypothesize that the pain induced by the conventional method inclusive preoperational lidocaine injection will be the same or more intense than using DNTT without local anesthesia. Secondly the investigators hypothesize that the use of DNTT for the placement of the arterial catheter will decrease the time spend, amount of complications (hematoma), the number of pricks, the number of utilized catheters compared to the traditional palpation method. Thirdly the investigators claim that the best anatomical place to put the catheter isn't always corresponding with the spot chosen by palpation, which increase the number of failures.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-90 years
* Fulfill the criteria of an operation
* Routine need of an arterial needle

Exclusion Criteria:

* Lack of patient consent
* Ultrasound identified plaques in the radial artery or ultrasound verified positive Allens test or traditional positive Allens test

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain score on visual analog scale | 5 minutes
  The primary outcome is the subjective feeling of pain following the two methods.

SECONDARY OUTCOMES:
Time spend on the procedure | 1 day
  Time will be measured from the point where 1) the operator starts searching for the patients plus or 2) the operator starts examining the patient with the ultrasound machine. The time will be stopped at the time where the catheter is successfully placed.
Number of utilized needles | 1 day
number of pricks | 1 day
  a prick is defined as eruption of the skin
number of withdrawals | 1 day
  a withdrawal is defined as backwards movement of the needle or the needle+catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Aa Hansen, stud.med, Principal Investigator — University of Aarhus
Locations (1):
- Anæstesiologisk-Intensiv afdeling I, Aarhus, Jylland, Denmark

REFERENCES:
- See also: Aarhus university Hospital, Skejby — http://www.auh.dk
- See also: The danish local ethical komité — http://www.komite.rm.dk